CLINICAL TRIAL: NCT05953168
Title: An Open-label, Single-arm Phase II Trial of First-line Treatment With Trastuzumab Deruxtecan for Patients With Locally Advanced or Metastatic Triple-Negative Breast Cancer, Luminal Androgen Receptor Subtype With Low Human Epidermal Growth Factor Receptor 2 (HER2) Expression.
Brief Title: T-DXd in the First-Line Treatment of Locally Advanced or Metastatic TNBC-LAR HER2-low Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N059
Record Dates: First submitted 2023-07-12; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Triple-Negative Breast Cancer
Keywords: triple-negative breast cancer; T-DXd treatment
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trastuzumab Deruxtecan (T-DXd) (Experimental)
  Interventions: Drug: Trastuzumab Deruxtecan

INTERVENTIONS:
Drug: Trastuzumab Deruxtecan — Trastuzumab Deruxtecan for TNBC-LAR patients with HER2 low expression

SUMMARY:
This is an open-label, single-arm phase II trial of first-line treatment with trastuzumab deruxtecan (T-DXd) for patients with locally advanced or metastatic triple-negative breast cancer, luminal androgen receptor subtype (TNBC-LAR) with low HER2 expression.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-70 years old;
2. Eastern Cooperative Oncology Group (ECOG) Performance Status Scale score 0 or 1;
3. Expected lifetime of not less than three months;
4. Disease-free interval >6 months；
5. Adequate tumor tissue samples collected within a time frame of less than 3 months;
6. Histological results recorded as TNBC [negative HER2, ER, and progesterone receptor (PgR) status] and LAR subtype according to the classification of Fudan University Shanghai Cancer Center (FUSCC);
7. Measurable disease according to Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1);
8. Cancer stage: recurrent or metastatic breast cancer; Local recurrence be confirmed by the researchers could not be radical resected;
9. Adequate hematologic and end-organ function, laboratory test results;
10. Within the 3 weeks prior to study initiation, patients have not received radiotherapy, endocrine therapy, targeted therapy, or surgery, and have recovered from acute toxicities associated with previous treatments (if surgery was performed, wound healing is complete); no peripheral neuropathy or grade I peripheral neurotoxicity.
11. Female subjects with fertility are required to use a medically approved contraceptive method during the study treatment；
12. Participants voluntarily joined the study, has signed informed consent before any trial related activities are conducted, has good compliance and has agreed to follow-up.

Exclusion Criteria:

1. Use of radiotherapy (except for palliative reasons), chemotherapy, and immunotherapy in the 3 weeks prior to treatment, excluding bisphosphonates (which can be used for bone metastasis)；
2. History of clinically uncontrolled heart disease, including congestive heart failure, angina, myocardial infarction within the past 6 months, or ventricular arrhythmias；
3. Common Terminology Criteria for Adverse Events (CTCAE) grade ≥1 adverse reactions attributed to previous treatments；
4. Underwent major surgery (excluding outpatient minor procedures, such as placement of vascular access) within the first 3 weeks of the investigational treatment；
5. Pregnant or lactating patients；
6. History of malignancy within the past five years (excluding cured basal cell carcinoma and cervical carcinoma in situ)；
7. Presence of third-space fluid accumulation (such as significant pleural effusion and ascites) that cannot be controlled by drainage or other methods；
8. Non-infectious interstitial lung disease (ILD) or non-infectious pneumonia requiring steroid hormone therapy, current ILD/non-infectious pneumonia, or suspected ILD/non-infectious pneumonia that cannot be ruled out by imaging examinations during screening (Note: Subjects found to have ILD/non-infectious pneumonia during baseline screening chest CT are ineligible)；
9. Known active Hepatitis B virus (HBV) or Hepatitis C virus (HCV) infection or HBV DNA ≥500, or patients with chronic phase accompanied by abnormal liver function；
10. Individuals with allergies or a history of known allergy to components of the study drugs or other monoclonal antibodies；
11. History of immunodeficiency, including HIV-positive test results, acquired or congenital immunodeficiency diseases, or history of organ transplantation. Positive syphilis antibody test；
12. According to the investigator's judgment, any evidence of diseases that the investigator considers unfavorable for the subject's participation in the study or that may affect their adherence to the protocol.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Objective Response of Complete Response (ORR) | 3 years (assessed at Screening, every 6 weeks for the first 12 months, thereafter every 9 weeks until disease progression or death, whichever occurs first)
  Percentage of Participants With an Objective Response of Complete Response (CR) or Partial Response (PR) According to Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 in all Participants

SECONDARY OUTCOMES:
Duration of response (DOR) | 3 years (assessed at Screening, every 6 weeks for the first 12 months, thereafter every 9 weeks until disease progression or death, whichever occurs first)
  Length of time that a tumor continues to respond to treatment without the cancer Duration of response is the time from response to progression/death
Disease Control Rate (DCR) | 3 years (assessed at Screening, every 6 weeks for the first 12 months, thereafter every 9 weeks until disease progression or death, whichever occurs first)
  Proportion of all subjects receiving study therapy whose best overall response is complete response (CR), partial response (PR), and stable disease (SD) for 8 weeks or more according to RECIST v1.1 criteria.
Progression Free Survival (PFS) | 3 years (assessed at Screening, every 6 weeks for the first 12 months, thereafter every 9 weeks until disease progression or death, whichever occurs first)
  Defined as the date from enrollment to the first recording of tumor progression (as measured by RECIST v1.1 criteria with or without continued treatment) or the date of death from any cause, whichever occurs first.
Overall Survival (OS) | Every 6 months
  Defined as the time from enrollment to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Breast cancer institute of Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided